CLINICAL TRIAL: NCT04977479
Title: A Randomized, Placebo-controlled Crossover Study to Assess the Safety of Administering a Second Dose of a COVID-19 mRNA Vaccine in Individuals Who Experienced a Systemic Allergic Reaction to an Initial Dose
Brief Title: The Safety of Administering a Second Dose of a COVID-19 mRNA Vaccine in Individuals Who Experienced a Systemic Allergic Reaction to an Initial Dose
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 10000460; 000460-I
Record Dates: First submitted 2021-07-24; First posted 2021-07-27 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-01

CONDITIONS: Systemic Allergic Reaction
Keywords: polyethylene glycol (PEG); Pfizer-BioNTech COVID-19 vaccine; Moderna Covid-19 vaccine; Consortium for Food Allergy Research (CoFAR); SARS-CoV-2; Comirnaty
MeSH Terms: interventions — BNT162 Vaccine; BNT162b5

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Blinded Active Vaccine 2 (Active Comparator): Participants who experienced a systemic allergic reaction after receiving their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine receives one dose of the active mRNA COVID-19 vaccine (0.3mL) intramuscularly followed by a wash out period of 24 hours then crossover to receive placebo (0.3 mL normal saline) intramuscularly.
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine (Comirnaty); Other: Placebo
- Blinded Placebo (Placebo Comparator): Participants who experienced a systemic allergic reaction after receiving their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine receives one dose of the placebo (0.3 mL normal saline) intramuscularly followed by a wash out period of 24 hours then crossover to receive the active mRNA COVID-19 vaccine (0.3mL) intramuscularly.
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine (Comirnaty); Other: Placebo
- Open-Label Booster Vaccine (Experimental): Participants who did not suffer from a COFAR grade 3 or higher reaction after blinded active vaccine 2 were offered to receive booster dose of the active mRNA COVID-19 vaccine (0.3 mL) intramuscularly 5 months later.
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine (Comirnaty); Biological: Pfizer-BioNTech COVID-19 Vaccine, Bivalent

INTERVENTIONS:
Biological: Pfizer-BioNTech COVID-19 Vaccine (Comirnaty) — mRNA vaccine for the prevention of COVID-19. Single dose (0.3mL) via IM.
Other: Placebo — Commercially available sterile, preservative-free 0.9% Sodium Chloride Injection, USP. Volume to match active vaccine controlling for and delivered as a single dose via IM.
  Arms: Blinded Active Vaccine 2; Blinded Placebo
Biological: Pfizer-BioNTech COVID-19 Vaccine, Bivalent — mRNA vaccine booster bivalent (Original and Omicron BA.4/BA.5) for the prevention of COVID-19. Single dose (0.3mL) via IM.
  Arms: Open-Label Booster Vaccine

SUMMARY:
Background:

Some people have allergic reactions to COVID-19 mRNA vaccines. Researchers want to learn more about these reactions to provide guidance on who can safely receive the vaccines, including a second dose in people who had a reaction to the first.

Objective:

To study the safety of giving a second mRNA COVID-19 vaccine dose to people who had a systemic allergic reaction to their first dose.

Eligibility:

People aged 16-69 who had a systemic allergic reaction to their first dose of COVID-19 vaccine.

Design:

Individuals who have underlying health issues may need to come to the NIH for screening tests to make sure they are safe to receive the vaccine. People who are eligible to participate in the study will be admitted to the NIH hospital and stay for at least 4 days. They will give urine samples. They will have a nasal swab SARS-CoV-2 test. They will have an intravenous line placed in each arm. They will get the study vaccine (Pfizer-BioNTech COVID-19 vaccine) and one dose of placebo on different days. They will have breathing tests. They may have clinical photography if they develop a rash.

Participants will have 4 follow-up visits - 2 by phone and 2 in-person visits at the NIH campus . They will have allergy skin testing at one visit. Drops of different allergens or controls will be placed on their back or arm. The skin under each drop will be scratched with a tool. If the results are negative, a small amount of allergen will be injected just below the surface of their skin. Participants who have no or only a mild allergic reaction to the second dose of the vaccine may be eligible to receive a Booster dose at the NIH.

Participation will last for approximately 5 months.

DETAILED DESCRIPTION:
Study Description:

This is a single-site study to determine the safety of administering a dose of the Pfizer-BioNTech mRNA coronavirus disease 2019 (COVID-19) vaccine (Comirnaty) to individuals who experienced a systemic allergic reaction to their first full dose of the same vaccine or the Moderna mRNA vaccine, and to investigate possible mechanisms underlying allergic reactions.

Objectives:

Primary Objective:

1. Assess the proportion of participants who develop a systemic allergic reaction (Consortium for Food Allergy Research grade 2 reaction and above regardless of tryptase, or CoFAR grade 1 with elevated tryptase [1.2 X baseline plus 2ng/mL]) to the Pfizer-BioNTech COVID-19 vaccine after previously demonstrating a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the same vaccine or the Moderna COVID-19 vaccine.

Secondary Objectives:

1. Assess the proportion of participants who develop a severe systemic allergic reaction (CoFAR Grade 3 reaction or higher regardless of tryptase) to the Pfizer-BioNTech COVID-19 vaccine after previously demonstrating a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the same vaccine or the Moderna COVID-19 vaccine.
2. Assess the proportion of participants who develop a mild-moderate allergic reaction (CoFAR Grade 1 or 2 reaction regardless of tryptase) to the Pfizer-BioNTech COVID-19 vaccine after previously demonstrating a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the same vaccine or the Moderna COVID-19 vaccine.
3. Assess the proportion of participants with anaphylactic reactions (Levels 1-3) per Brighton Collaboration Criteria (see Appendix B) to the Pfizer-BioNTech COVID-19 vaccine after previously demonstrating a systemic allergic reaction (CoFAR Grade 2 or 3 reaction OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the same vaccine or the Moderna COVID-19 vaccine.
4. Assess the proportion of participants who develop a systemic allergic reaction (CoFAR Grade 2 reaction or higher regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to the Pfizer-BioNTech COVID-19 vaccine after previously demonstrating a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the same vaccine or the Moderna COVID-19 vaccine compared to the rate of these reactions following placebo administration.
5. Compare the severity of allergic reactions to the first dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine to the severity of the reaction following administration of a subsequent dose of the Pfizer-BioNTech vaccine in individuals who experienced a systemic allergic reaction (CoFAR grade 2 reaction and above regardless of tryptase, or CoFAR grade 1 with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine.

Exploratory Objectives:

1. Assess the risk of having a systemic allergic reaction to a dose of the Pfizer-BioNTech COVID-19 vaccine in participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the same vaccine or the Moderna COVID-19 according to baseline covariates.
2. Examine possible mechanisms of allergic reactions to mRNA-based COVID-19 vaccines.
3. Assess innate and adaptive immune responses, including functional antibody levels, to the Pfizer-BioNTech COVID-19 vaccine
4. Investigate mental health characteristics of participants who experience an allergic reaction to the COVID-19 vaccine.
5. Assess psychological impact of allergic reactions to the COVID-19 vaccine and examine changes in stress levels over time.
6. Assess anxiety levels in participants and examine changes in anxiety over time.
7. Assess the proportion of participants who experience no reaction or only a mild reaction (CoFAR Grade 2 or below) to a booster dose of the Pfizer-BioNTech vaccine after previously demonstrating a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2 ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine and no allergic reaction or a mild reaction (CoFAR Grade 2 or below) to a subsequent (second) dose of the Pfizer-BioNTech vaccine.
8. Assess the development of autoantibodies after COVID-19 vaccination.

Endpoints:<TAB>

Primary Endpoint:

1. The proportion of participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine who experience a systemic allergic reaction (CoFAR Grade 2 and above reaction regardless of tryptase, or CoFAR grade 1 with elevated tryptase [1.2 X baseline plus 2ng/mL]) within the 3-hour post-vaccine observation period to a subsequent dose of the Pfizer-BioNTech vaccine.

Secondary Endpoints:

1. The proportion of participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine who experience a severe systemic allergic reaction (CoFAR grade 3 reaction and above) within the 3-hour post-vaccine observation period to a subsequent dose of the Pfizer-BioNTech vaccine.
2. The proportion of participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine who experience a mild-moderate allergic reaction (CoFAR grade 1 or 2 reaction regardless of tryptase) within the 3-hour post-vaccine observation period to a subsequent dose of the Pfizer-BioNTech vaccine.
3. The proportion of participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine who experience an anaphylactic reaction (Levels 1-3) per Brighton Collaboration Criteria within the 3-hour post-vaccine observation period to a subsequent dose of the Pfizer-BioNTech vaccine.
4. The proportion of participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine who experience a systemic allergic reaction (CoFAR grade 2 reaction and above regardless of tryptase, or CoFAR grade 1 with elevated tryptase [1.2 X baseline plus 2ng/mL]) within the 3-hour post-vaccine observation period to a subsequent dose of the Pfizer-BioNTech vaccine compared to the rate of these reactions following placebo administration.
5. The proportion of participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine who develop a lower or higher grade allergic reaction within the 3-hour post-vaccine observation period to a subsequent dose of the Pfizer-BioNTech vaccine.

Exploratory Endpoints:

1. Prevalence of polyethylene glycol (PEG) and severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) antibodies in each participant at baseline.
2. Changes in anti-PEG and SARS-CoV-2 antibodies in each participant approximately 1 and 5 months after receiving the dose of the Pfizer-BioNTech vaccine administered on study.
3. Prevalence of positive skin testing to the vaccine and/or vaccine components including PEG- and polysorbate 80-containing medications.
4. Changes in biomarkers from baseline to post-dose of the Pfizer-BioNTech vaccine administered on study (e.g., known mediators of systemic reactions due to mast cell activation, markers of inflammatory response, markers of basophil and neutrophil activation, markers associated with activation of the classical and alternative complement pathways or kinin system, proteomics, metabolomics).
5. Changes in blood transcriptomics after vaccination.
6. Changes in innate and adaptive immune responses including functional antibody levels after vaccination.
7. Mental health/anxiety questionnaire scores and anxiety level ratings at baseline.
8. Results of psychiatric consultation/mental health interview.
9. Changes in mental health/anxiety questionnaire scores and anxiety level ratings over the study period.
10. The proportion of participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2 ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine and no allergic reaction or a mild reaction (CoFAR Grade 2 or below) to a subsequent (second) dose of the Pfizer-BioNTech vaccine who experience no reaction or only a mild reaction (CoFAR Grade 2 or below) to a booster dose of the Pfizer-BioNTech vaccine administered approximately 5 months after the second dose.
11. Changes in blood transcriptomics after vaccination.
12. Changes in innate and adaptive immune responses including functional antibody levels after vaccination.
13. Mental health/anxiety questionnaire scores and anxiety level ratings at baseline.
14. Results of psychiatric consultation/mental health interview.
15. Changes in mental health/anxiety questionnaire scores and anxiety level ratings over the study period.
16. The proportion of participants who previously demonstrated a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless

    of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2 ng/mL]) to their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine and no allergic reaction or a mild reaction (CoFAR Grade 2 or below) to a subsequent (second) dose of the Pfizer-BioNTech vaccine who experience no reaction or only a mild reaction (CoFAR Grade 2 or below) to a booster dose of the Pfizer-BioNTech vaccine administered approximately 5 months after the second dose.
17. The development of autoantibodies post-second and post-booster doses of the COVID-19 mRNA vaccines.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Ability to provide informed consent.
* Stated willingness to comply with all study procedures (including discontinuing medications as needed and availability for the duration of the study.
* Aged 16-69 years.
* Must have experienced a systemic allergic reaction (CoFAR Grade 2 or 3 reaction regardless of tryptase OR Grade 1 reaction with elevated tryptase [1.2 X baseline plus 2 ng/mL] per modified CoFAR Grading Scale for Systemic Allergic Reactions Version 3.0) to the first dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine. Patients without documented hypoxia, hypotension, or evidence of end-organ damage who were treated with epinephrine infusion would be considered as CoFAR Grade 3 reaction and may be eligible per investigator discretion.
* Must be at least 28 days out from their first dose of the Moderna vaccine or 21 days from their first dose of the Pfizer-BioNTech vaccine before proceeding with the placebo or vaccine challenge in this study.
* Have a primary care physician or other health care provider who will manage their medical care outside of this study.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Experienced a Grade 4 systemic allergic reaction (per CoFAR Grading Scale for Systemic Allergic Reactions Version 3.0) to the first dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine.
* Known exposure to SARS-CoV-2 and still within the quarantine window.
* Symptoms consistent with acute COVID-19 infection or known COVID-19 infection (positive reverse transcription-polymerase chain reaction [RT-PCR] or antigen test) and still within the quarantine window
* Have an acute illness, including body temperature greater than 100.4 degrees F, within 14 days prior to enrollment.
* History of autoimmune or other disorders requiring systemic immune modulators.
* Are moderately or severely immunocompromised.
* History of acute urticaria within 28 days prior to enrollment.
* Pregnant.
* Have received any vaccines within 14 days prior to enrollment.
* Scheduled or planned receipt of approved or experimental vaccine prior to visit 3.
* Had any allergen immunotherapy administration within 24 hours prior to the first study vaccination or plan to receive within 24 hours after the second study vaccination.
* Have received a biological therapy within 6 months prior to enrollment.
* Use of systemic steroids for any reason within 28 days prior to enrollment.
* Use of zileuton within 14 days prior to enrollment.
* Use of EUA monoclonal antibodies casirivimab and indevimab, or bamlanivimab, or any other antibody agent for treatment or prevention of COVID-19 within 3 months of randomization.
* Presence of condition(s) that, in the judgment of the investigator or the referring physician, may put the participant at undue risk or make them unsuitable for participation in the study.

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela A Guerrerio, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Kee SA, Olivera A, Chatman L, Khalid MB, Li MJ, Chu E, Zektser E, Laky K, Frischmeyer-Guerrerio PA. Basophil activation test to BNT162b2 lacks specificity for predicting allergic reactions to the mRNA vaccine. J Allergy Clin Immunol Glob. 2025 May 13;4(3):100495. doi: 10.1016/j.jacig.2025.100495. eCollection 2025 Aug. PMID 40497015
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000460-I.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants withdrew prior to start of study. One participant was ineligible due to partial 2nd vaccine dose pre-enrollment outside of the study
Period: First Period of Crossover
Arm/Group | Blinded Active Vaccine 2 | Blinded Placebo | Open-Label Booster Vaccine
Started | 8 | 8 | 0
Completed | 8 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Blinded Active Vaccine 2 | Blinded Placebo | Open-Label Booster Vaccine
Started | 8 | 8 | 0
Completed | 8 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Second Period of Crossover
Arm/Group | Blinded Active Vaccine 2 | Blinded Placebo | Open-Label Booster Vaccine
Started | 8 | 8 | 0
Completed | 8 | 8 | 0
Not Completed | 0 | 0 | 0
Period: Open Label
Arm/Group | Blinded Active Vaccine 2 | Blinded Placebo | Open-Label Booster Vaccine
Started | 0 | 0 | 16
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinded Active Vaccine 2 | Blinded Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Had Recurrent Systemic Allergic Reaction to Vaccine
Description: Proportion of participants who had recurrent systemic allergic reaction following active COVID-19 vaccine dose in this study. Allergic reactions were graded using Consortium of Food Allergy Research (CoFAR) grading scale (Version 3.0) where Grade 1 (mild) = mild symptoms involving one organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 2 (moderate) = mild symptoms involving ≥2 organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 3 (severe)= moderate to severe cardiovascular, lower respiratory or gastrointestinal symptoms, responsive to treatment and/or without end-organ dysfunction; Grade 4 = severe cardiovascular or lower respiratory symptoms, with end-organ dysfunction and/or refractory to treatment; and Grade 5 = death.
  Systemic allergic reaction was defined as CoFAR grade 1 reaction with elevated tryptase or CoFAR Grade ≥ 2 reaction irrespective of tryptase levels.
Time Frame: Within the 3-hour post-vaccine observation period
Population: The analysis included participants who received the active study vaccine in the crossover phase as pre-specified in the protocol to only collect and report data from the active vaccination.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Blinded Active Vaccine 2: Participants who experienced a systemic allergic reaction after receiving their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine receives one dose of the active mRNA COVID-19 vaccine (0.3mL) intramuscularly
Arm/Group | Blinded Active Vaccine 2
Number analyzed (Participants) | 16
Proportion of participants | 0.125 [0.016 to 0.383]

2. Primary Outcome: Proportion of Participants Who Had Recurrent Systemic Allergic Reaction to Vaccine
Description: as for outcome 1
Time Frame: Within the 3-hour post-vaccine observation period
Population: The analysis included participants who received both active study vaccines in the crossover phase and the booster dose in the open label phase
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Open-Label Booster Vaccine
Number analyzed (Participants) | 16
Proportion of participants | 0.125 [0.016 to 0.383]

3. Secondary Outcome: Proportion of Participants Who Developed Severe Systemic Allergic Reaction to Vaccine
Description: Proportion of participants who developed severe systemic allergic reaction following active COVID-19 vaccine dose in this study. Allergic reactions were graded using Consortium of Food Allergy Research (CoFAR) grading scale (Version 3.0) where
  Grade 1 (mild) = mild symptoms involving one organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 2 (moderate) = mild symptoms involving ≥2 organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 3 (severe)= moderate to severe cardiovascular, lower respiratory or gastrointestinal symptoms, responsive to treatment and/or without end-organ dysfunction; Grade 4 = severe cardiovascular or lower respiratory symptoms, with end-organ dysfunction and/or refractory to treatment; and Grade 5 = death.
  Severe systemic allergic reaction was defined as CoFAR Grade ≥ 3 reaction, regardless of tryptase levels.
Time Frame: Within the 3-hour post-vaccine observation period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Blinded Active Vaccine 2
Number analyzed (Participants) | 16
Proportion of participants | 0 [0 to 0.206]

4. Secondary Outcome: Proportion of Participants Who Developed Severe Systemic Allergic Reaction to Vaccine
Description: as for outcome 3
Time Frame: Within the 3-hour post-vaccine observation period
Population: The analysis included those who had a systemic allergic reaction following 1st dose of an mRNA vaccine before study and received both active study active vaccines
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Open-Label Booster Vaccine
Number analyzed (Participants) | 16
Proportion of participants | 0.062 [0.002 to 0.302]

5. Secondary Outcome: Proportion of Participants Who Developed Mild or Moderate Systemic Allergic Reaction Following Active Vaccine Dose
Description: Proportion of participants who developed mild or moderate systemic allergic reaction following active COVID-19 vaccine dose in this study. Allergic reactions were graded using Consortium of Food Allergy Research (CoFAR) grading scale (Version 3.0) where
  Grade 1 (mild) = mild symptoms involving one organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 2 (moderate) = mild symptoms involving ≥2 organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 3 (severe)= moderate to severe cardiovascular, lower respiratory or gastrointestinal symptoms, responsive to treatment and/or without end-organ dysfunction; Grade 4 = severe cardiovascular or lower respiratory symptoms, with end-organ dysfunction and/or refractory to treatment; and Grade 5 = death
  Mild to moderate systemic allergic reaction was defined as CoFAR Grade 1 or 2 regardless of tryptase level.
Time Frame: Within the 3-hour post-vaccine observation period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Blinded Active Vaccine 2
Number analyzed (Participants) | 16
Proportion of participants | 0.188 [0.04 to 0.456]

6. Secondary Outcome: Proportion of Participants Who Developed Mild or Moderate Systemic Allergic Reaction Following Active Vaccine Dose
Description: Proportion of participants who had recurrent systemic allergic reaction following active COVID-19 vaccine dose in this study. Allergic reactions were graded using Consortium of Food Allergy Research (CoFAR) grading scale (Version 3.0) where grade 1 (mild) = mild symptoms involving one organ system (skin, conjunctiva, upper respiratory or gastrointestinal); grade 2 (moderate) = mild symptoms involving =2 organ system (skin, conjunctiva, upper respiratory or gastrointestinal); grade 3 (severe)= moderate to severe cardiovascular, lower respiratory or gastrointestinal symptoms, responsive to tr
Time Frame: Within the 3-hour post-vaccine observation period
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Open-Label Booster Vaccine
Number analyzed (Participants) | 16
Proportion of participants | 0.062 [0.002 to 0.302]

7. Secondary Outcome: Proportion of Participants Who Developed Anaphylactic Reaction Following Active Dose Delivered
Description: Proportion of participants with anaphylactic reactions (Levels 1-3) per Brighton Collaboration Criteria to the COVID-19 vaccine after previously demonstrating a systemic allergic reaction to their first full dose of the COVID-19 vaccine. Anaphylaxis was defined using the Brighton Collaboration Criteria as a clinical syndrome characterized by a sudden onset and rapid progression of signs and symptoms involving ≥2 organ systems including skin, cardiovascular, respiratory, gastrointestinal or tryptase elevation (>upper normal limit). Only specific clinical features from these organ systems meet major and/or minor criteria to provide level of diagnostic certainty for anaphylactic reaction. Reaction meeting levels 1-3 diagnostic certainty are consistent with anaphylaxis
Time Frame: Within the 3-hour post-vaccine observation period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Blinded Active Vaccine 2
Number analyzed (Participants) | 16
Proportion of participants | 0.062 [0.002 to 0.302]

8. Secondary Outcome: Proportion of Participants Who Developed Anaphylactic Reaction Following Active Vaccine Dose
Description: as for outcome 7
Time Frame: Within the 3-hour post-vaccine observation period
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Open-Label Booster Vaccine
Number analyzed (Participants) | 16
Proportion of participants | 0.062 [0.002 to 0.302]

9. Secondary Outcome: Proportion of Participants Who Had Recurrent Systemic Allergic Reaction Following Active Vaccine Dose Compared With Rate of Reaction in Placebo
Description: Participants with recurrent systemic allergic reaction following active vaccine dose in this study compared with reaction in placebo. Allergic reactions were graded using Consortium of Food Allergy Research (CoFAR) grading scale (Version 3.0) where Grade 1 (mild)= mild symptoms involving one organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 2 (moderate)= mild symptoms involving ≥2 organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 3 (severe)= moderate to severe cardiovascular, lower respiratory or gastrointestinal symptoms, responsive to treatment and/or without end-organ dysfunction; Grade 4= severe cardiovascular or lower respiratory symptoms, with end-organ dysfunction and/or refractory to treatment; and Grade 5= death Systemic allergic reaction was defined as CoFAR grade 1 reaction with elevated tryptase or CoFAR Grade ≥ 2 reaction irrespective of tryptase level. Outcome was calculated as risk difference estimation.
Time Frame: Within the 3-hour post-vaccine observation period
Population: The analysis included the proportion of participants who had a systemic allergic reaction after receiving the active study vaccine compared to the proportion who had a systemic allergic reaction after receiving placebo during the crossover phase of the study.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Blinded Active Vaccine 2: Participants who experienced a systemic allergic reaction after receiving their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine receives one dose of the active mRNA COVID-19 vaccine (0.3mL) intramuscularly in the crossover phase of the study.
- Placebo: Participants who experienced a systemic allergic reaction after receiving their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine receives one dose placebo (0.3 mL normal saline) intramuscularly in the crossover phase of the study.
Arm/Group | Blinded Active Vaccine 2 | Placebo
Number analyzed (Participants) | 16 | 16
Proportion of participants | 0.125 [-0.134 to 0.383] | 0 [0 to 0]

10. Secondary Outcome: Proportion of Participants With Less Severe Allergic Reaction to the Vaccine Dose Delivered in This Study Than Recorded Reaction to the First Full COVID-19 Vaccine Dose
Description: Proportion of participants with less severe allergic reaction to the vaccine dose in this study than recorded reaction to the first full COVID-19 vaccine dose (pre-study). Allergic reactions were graded using Consortium of Food Allergy Research (CoFAR) grading scale (Version 3.0) where
  Grade 1 (mild) = mild symptoms involving one organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 2 (moderate) = mild symptoms involving ≥2 organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 3 (severe)= moderate to severe cardiovascular, lower respiratory or gastrointestinal symptoms, responsive to treatment and/or without end-organ dysfunction; Grade 4 = severe cardiovascular or lower respiratory symptoms, with end-organ dysfunction and/or refractory to treatment; and Grade 5 = death.
  Systemic allergic reaction was defined as CoFAR grade 1 reaction with elevated tryptase or CoFAR Grade ≥ 2 reaction irrespective of tryptase levels.
Time Frame: Within the 3-hour post-vaccine observation period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Blinded Active Vaccine 2
Number analyzed (Participants) | 16
Proportion of participants | 0.188 [0.04 to 0.456]

11. Secondary Outcome: Proportion of Participants With Less Severe Allergic Reaction to the Vaccine Dose Delivered in This Study Than Recorded Reaction to the First Full COVID-19 Vaccine Dose
Description: as for outcome 10
Time Frame: Within the 3-hour post-vaccine observation period
Population: The analysis included those who had a systemic allergic reaction following 1st dose of an mRNA vaccine before study and received both active study active vaccines (blinded and open-label)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Open-Label Booster Vaccine
Number analyzed (Participants) | 16
Proportion of participants | 0.062 [0.002 to 0.302]

12. Secondary Outcome: Proportion of Participants With More Severe Systemic Allergic Reaction to the Vaccine Dose Delivered in This Study Than Recorded Reaction to the First Full Vaccine Dose
Description: "Proportion of participants with more severe allergic reaction to the vaccine dose in this study than recorded reaction to the first full COVID-19 vaccine dose (pre-study). Allergic reactions were graded using Consortium of Food Allergy Research (CoFAR) grading scale (Version 3.0) where
  Grade 1 (mild) = mild symptoms involving one organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 2 (moderate) = mild symptoms involving ≥2 organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 3 (severe)= moderate to severe cardiovascular, lower respiratory or gastrointestinal symptoms, responsive to treatment and/or without end-organ dysfunction; Grade 4 = severe cardiovascular or lower respiratory symptoms, with end-organ dysfunction and/or refractory to treatment; and Grade 5 = death
  Systemic allergic reaction was defined as CoFAR grade 1 reaction with elevated tryptase or CoFAR Grade ≥ 2 reaction irrespective of tryptase levels.
Time Frame: Within the 3-hour post-vaccine observation period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Blinded Active Vaccine 2
Number analyzed (Participants) | 16
Proportion of participants | 0 [0 to 0.206]

13. Secondary Outcome: Proportion of Participants With More Severe Systemic Allergic Reaction to the Vaccine Dose Delivered in This Study Than Recorded Reaction to the First Full Vaccine Dose
Description: "Proportion of participants with more severe allergic reaction to the vaccine dose in this study than recorded reaction to the first full COVID-19 vaccine dose (pre-study). Allergic reactions were graded using Consortium of Food Allergy Research (CoFAR) grading scale (Version 3.0) where
  Grade 1 (mild) = mild symptoms involving one organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 2 (moderate) = mild symptoms involving ≥2 organ system (skin, conjunctiva, upper respiratory or gastrointestinal); Grade 3 (severe)= moderate to severe cardiovascular, lower respiratory or gastrointestinal symptoms, responsive to treatment and/or without end-organ dysfunction; Grade 4 = severe cardiovascular or lower respiratory symptoms, with end-organ dysfunction and/or refractory to treatment; and Grade 5 = death.
  Systemic allergic reaction was defined as CoFAR grade 1 reaction with elevated tryptase or CoFAR Grade ≥ 2 reaction irrespective of tryptase levels.
Time Frame: Within the 3-hour post-vaccine observation period
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Open-Label Booster Vaccine
Number analyzed (Participants) | 16
Proportion of participants | 0 [0 to 0.206]

ADVERSE EVENTS:
Time Frame: Blinded Active Vaccine 2 & Placebo - Within 3-hour post-vaccination Overall Study - up to 17 months post intervention in the crossover phase Open-Label Booster Vaccine - up to 11 months post vaccine administration
Description: Adverse events associated with the crossover phase have been grouped under 'Overall Study' due to the brief washout period between the active vaccine and the placebo.
Groups:
- Placebo: Participants who experienced a systemic allergic reaction after receiving their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine receives one dose of placebo (0.3 mL normal saline) intramuscularly.
- Overall Study: Participants who experienced a systemic allergic reaction after receiving their first full dose of the Pfizer-BioNTech or Moderna COVID-19 vaccine receives one dose of the active mRNA COVID-19 vaccine (0.3mL) intramuscularly or placebo (0.3 mL normal saline) intramuscularly in the crossover phase of study.
Arm/Group | Blinded Active Vaccine 2 | Placebo | Open-Label Booster Vaccine | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 0/16 | 16/16 | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Active Vaccine 2 (N=16) | Placebo (N=16) | Open-Label Booster Vaccine (N=16) | Overall Study (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 (2) | 4 (5)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 | 0 | 4 (6) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 5 (5) | 8 (12)
Tachycardia (Cardiac disorders) | 0 | 0 | 1 (1) | 1 (2)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 | 0 | 1 (1) | 2 (3)
Lacrimation increased (Eye disorders) | 0 | 0 | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 | 0 | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 (4) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 3 (5)
Nausea (Gastrointestinal disorders) | 0 | 0 | 7 (9) | 8 (11)
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 0 | 0 | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 | 0 | 2 (2) | 6 (8)
Chest pain (General disorders) | 0 | 0 | 0 (0) | 1 (2)
Chills (General disorders) | 0 | 0 | 7 (8) | 8 (15)
Discomfort (General disorders) | 0 | 0 | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 | 0 | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 | 0 | 13 (15) | 12 (16)
Feeling abnormal (General disorders) | 0 | 0 | 1 (1) | 1 (1)
Feeling hot (General disorders) | 0 | 0 | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 | 0 | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 | 0 | 10 (14) | 8 (11)
Injection site induration (General disorders) | 0 | 0 | 9 (10) | 2 (3)
Injection site oedema (General disorders) | 0 | 0 | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 | 0 | 14 (15) | 14 (16)
Injection site pruritus (General disorders) | 0 | 0 | 2 (2) | 2 (2)
Injection site reaction (General disorders) | 0 | 0 | 0 (0) | 2 (2)
Injection site warmth (General disorders) | 0 | 0 | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 | 0 | 1 (1) | 1 (1)
Tenderness (General disorders) | 0 | 0 | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 | 0 | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 | 3 (3) | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 | 0 | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 | 0 | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 0 | 0 | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 | 0 | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 | 0 | 9 (9) | 11 (19)
Eosinophil count increased (Investigations) | 0 | 0 | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 (1) | 8 (9)
Lymphocyte count increased (Investigations) | 0 | 0 | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 | 0 | 0 (0) | 1 (2)
Neutrophil count increased (Investigations) | 0 | 0 | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 | 0 | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 | 0 | 0 (0) | 4 (4)
White blood cell count increased (Investigations) | 0 | 0 | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 (2) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 (4) | 6 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9 (9) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 | 0 | 6 (6) | 9 (12)
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 | 0 | 12 (14) | 12 (13)
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 (2) | 1 (2)
Migraine (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 | 0 | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 | 0 | 6 (6) | 7 (9)
Parosmia (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 | 0 | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 | 0 | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 0 | 0 | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 (0) | 1 (1)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 2 (3)
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 (6) | 4 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 (4) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 (3) | 2 (3)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 (4) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 (7) | 6 (7)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 (4) | 4 (4)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 (3) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 (2) | 3 (3)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (2) | 10 (17)
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 (3) | 3 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 1 (1)
Bereavement (Social circumstances) | 0 | 0 | 1 (1) | 0 (0)
Catheter management (Surgical and medical procedures) | 0 | 0 | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 | 0 | 2 (3) | 3 (4)
Haematoma (Vascular disorders) | 0 | 0 | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 | 0 | 1 (1) | 3 (5)
Hypotension (Vascular disorders) | 0 | 0 | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There was no pre-determined method for addressing causality of adverse events in the crossover phase of the study due to the brief washout period between the active vaccine and placebo administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT04977479/Prot_SAP_000.pdf